CLINICAL TRIAL: NCT04021433
Title: Ketamine for Treatment Resistant Depression - A Long Term Feasibility Study
Brief Title: Ketamine for Treatment Resistant MDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 58717-HMO-CTIL
Record Dates: First submitted 2019-07-10; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MDD (Experimental): Treatment resistant patients will be treated with multiple doses of IM/SC ketamine [dose range 0.3-1.5mg/kg]
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Repeated doses of IM/SC ketamine up to 3 times a week

SUMMARY:
This study aims to openly test the long-term safety, tolerability and effectiveness of repeated administration of IM/SC ketamine for treatment resistant MDD.

DETAILED DESCRIPTION:
Major depression disorder (MDD) is a common psychiatric disorders with considerable impact on patients' quality of life, social and occupational function. MDD also significantly increase suicide rate. About a third of the patients with MDD suffer from moderate to severe symptoms that are fully or partially unresponsive to accepted pharmaco and / or psycho therapy. Ketamine is a widely used anesthetic. Multiple studies done over the recent years had shown its therapeutic effects in resistant depressive patients. Unlike regular antidepressants, ketamine exerts its effect within hours to few days which implies an alternative mechanism of action not fully studied. So far, there are only few reports on using repeated ketamine administration to maintain the antidepressant effect or on intra-muscular or sub-cutaneous application that can be safer and more tolerable than the intravenous route.

In the present study, the investigators aim to openly assess the safety, tolerability and effectiveness of repeated, individually tailored IM or SC ketamine for treatment resistant major depression. The investigators intend to explore questions regarding optimal dose, treatment frequency and duration. The investigators will also assess potential cognitive effects of long-term ketamine treatment and look for possible treatment outcome predictors using the Neurotrax computerized cognitive battery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with unipolar/bipolar depression with MADRS Score>= 20
* Inadequate response to >= 3 adequate treatment trials [>=2 trials in the present episode]
* If on psychopharmacological Tx, it should be stable since 4 weeks prior to enrollment
* QTc WNL

Exclusion Criteria:

* Hypersensitivity to ketamine
* Other major psychiatric diagnosis
* High suicidality
* Unstable physical illness
* S/P CVA / brain SOL
* Pregnant or breast feeding women
* Illicit drug/alcohol abuse during last year
* History of ketamine abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
MADRS | 1 month into treatment through study completion
  The change in the MDRS score at 1 month (5weeks evaluation) for the acute phase and at 6 months or end of study (for the maintenance phase) compared to baseline

SECONDARY OUTCOMES:
MADRS | 3 months into treatment
  The change in MADRS score at 3 months compared to baseline.
QIDS-SR, Clinical Global Impressions - Improvement | along 6 months
  The change in QIDS-SR and CGI scores at 1, 3 and 6 months compared to baseline.
Average time in remission | along 6 months
  Average time in remission.
NeuroTrax computerized cognitive battery | along 6 months
  Changes in cognitive function at 1 and 6 months [or at study end] as assessed by the NeuroTrax computerized cognitive battery compared to baseline.
  correlation between information processing speed and other cognitive domains at baseline and clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel